CLINICAL TRIAL: NCT01688622
Title: Effects of Exercise on Glypican4,CTRP3,5 and RBP4 Levels and Circulating Levels of These Adipokines in the Subjects With or Without Metabolic Syndrome
Brief Title: Glypican4 and CTRP5 in Metabolic Syndrome and the Effect of Exercise on These Adipokines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, K. M. Choi, Professor, Korea University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: KoreaSO_Exercise
Record Dates: First submitted 2012-09-13; First posted 2012-09-20 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Metabolic Syndrome; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise (Other): obese women who are volunteers for the 3 months exercise programs
  Interventions: Behavioral: 3months Exercise

INTERVENTIONS:
Behavioral: 3months Exercise — training session consisting of a brief warm-up, followed by an approximately 45-min session of aerobic exercise at an intensity of 60-75% of the age-predicted maximum heart rate (approximately 300 kcal/day) and a 20-min muscle strength train- ing programme (approximately 100 kcal/day), followed by a brief cool-down period.

SUMMARY:
Glypican4, CTRP3, CTRP5 are emerging novel adipokines mediating obesity and inflammation related disorders. RBP4 and adiponectin are well known important adipokines. Therefore, we examine the circulating levels of theses adipokines in the subjects with or without metabolic syndrome. Furthermore, we tried to clarify the effect of exercise on the circulating these adipokines.

ELIGIBILITY:
Inclusion Criteria:

* Women between 30 and 60 years of age who had a body mass index (BMI) more than 25 kg/m2
* The subjects of metabolic syndrome and age, gender matched non metabolic syndrome among the participants of Korean SO Study (KSOS) study, which is an ongoing epidemiologic study supported by the Korea Science and Engineering Foundation

Exclusion Criteria:

* participants had a history of cardiovascular disease
* any type of diabetes
* stage 2 hypertension
* malignant disease, severe renal, or hepatic disease
* Subjects taking medications that might affect body weight or body composition

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The changes of circulating glypican4 levels after 3 months exercise | baseline and 12weeks
The changes of circulating CTRP3 levels after 3 months exercise | baseline and 12weeks
The changes of circulating CTRP5 levels after 3 months exercise | baseline and 12weeks
The changes of circulating RBP4 levels after 3 months exercise | baseline and 12weeks
The changes of circulating adiponectin levels after 3 months exercise | baseline and 12weeks

SECONDARY OUTCOMES:
Circulating glypican4 levels in the subjects with or without metabolic syndrome | baseline
Circulating CTRP3 levels in the subjects with or without metabolic syndrome | baseline
Circulating CTRP5 levels in the subjects with or without metabolic syndrome | baseline
Circulating RBP4 levels in the subjects with or without metabolic syndrome | baseline
Circulating adiponectin levels in the subjects with or without metabolic syndrome | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Choi HY, Park JW, Lee N, Hwang SY, Cho GJ, Hong HC, Yoo HJ, Hwang TG, Kim SM, Baik SH, Park KS, Youn BS, Choi KM. Effects of a combined aerobic and resistance exercise program on C1q/TNF-related protein-3 (CTRP-3) and CTRP-5 levels. Diabetes Care. 2013 Oct;36(10):3321-7. doi: 10.2337/dc13-0178. Epub 2013 Jun 18. PMID 23780948
- [Derived] Yoo HJ, Hwang SY, Cho GJ, Hong HC, Choi HY, Hwang TG, Kim SM, Bluher M, Youn BS, Baik SH, Choi KM. Association of glypican-4 with body fat distribution, insulin resistance, and nonalcoholic fatty liver disease. J Clin Endocrinol Metab. 2013 Jul;98(7):2897-901. doi: 10.1210/jc.2012-4297. Epub 2013 Apr 30. PMID 23633195